CLINICAL TRIAL: NCT06690229
Title: Evaluation of Different Cementation Materials Used in Prefabricated Pediatric Zirconia Crowns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Kadriye Görkem Ulu Güzel, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/037
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Caries,Dental
Keywords: Early childhood caries; Zirconia crown; Cementation
MeSH Terms: conditions — Dental Caries | interventions — Glass Ionomer Cements; Ketac-cem; RelyX U200

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glass ionomer cement (Experimental): Prefabricated zirconia crowns cemented with glass ionomer cement (Ketac Cem (3M ESPE, USA)) on primary maxillary incisors will be clinically evaluated at 1-week, 3-month, 6-month, and 12-month follow-ups in terms of periodontal health, plaque accumulation, wear of opposing teeth, parental satisfaction, color match, retention, marginal integrity, and contact harmony
  Interventions: Drug: glass ionomer cement
- dual-cure self-adhesive resin cement (Experimental): Prefabricated zirconia crowns will be cemented with dual-cure self-adhesive resin cement (RelyX U200 (3M ESPE, St. Paul, USA)) on primary maxillary incisors and will be evaluated during follow-up sessions.
  Interventions: Drug: self-adhesive resin cement
- resin modified glass ionomer cement (Experimental): Prefabricated zirconia crowns will be cemented with resin modified glass ionomer cement (FujiCEM Evolve (GC, Tokyo, Japan)) on primary maxillary incisors and will be evaluated during follow-up sessions.
  Interventions: Drug: resin modified glass ionomer cement

INTERVENTIONS:
Drug: glass ionomer cement — A cement used for crown cementation
  Other Names: Ketac Cem (3M ESPE, USA)
  Arms: glass ionomer cement
Drug: self-adhesive resin cement — A cement used for crown cementation
  Other Names: RelyX U200 (3M ESPE, St. Paul, USA)
  Arms: dual-cure self-adhesive resin cement
Drug: resin modified glass ionomer cement — A cement used for crown cementation
  Other Names: FujiCEM Evolve (GC, Tokyo, Japan)
  Arms: resin modified glass ionomer cement

SUMMARY:
Today, with increasing aesthetic demands; the need for materials that are both durable and compatible with the appearance of natural teeth is increasing in paediatric dentistry. Prefabricated zirconium crowns have attracted significant interest in recent years because they meet aesthetic expectations and have offer mechanical strength. There are various traditional and contemporary cement options that can be used for cementation of crowns.

The aim of this study is to clinically evaluate prefabricated zirconia crowns cemented to the primary maxillary incisors with three different adhesive cements in terms of periodantal health, plaque accumulation, opposing tooth wear, parental satisfaction, color harmony, retention, marginal integrity and contact compatibility, at the 1-week, 3-month, 6-month, 12-month follow-ups.

DETAILED DESCRIPTION:
The sample size was calculated as 30 with the G*Power analysis program. Considering the case losses, the sample size will be increased by 20% and a total of 36 teeth will be included. In the study, 3 different cements will be applied to each cement group, 12 teeth.

In this study, 36 teeth will be included from patients aged 3-4 years who have two or more surface carious lesions on their maxillary incisors. After necessary caries removal and pulpectomy treatment, prefabricated zirconia crowns will be prepared and cemented under general anesthesia, using one of three randomly selected cements.

12 teeth will be cemented with FujiCEM Evolve (GC, Tokyo, Japan) 12 teeth with RelyX U200 (3M ESPE, St. Paul, USA) 12 teeth with Ketac Cem (3M ESPE, USA) Patients will be called for follow-up examinations one week after the completion of all dental treatments and at 3, 6, and 12 months. During these follow-ups, Gingival Index, Plaque Index, Tooth Wear Index, and Ryge (USPHS) Criteria will be evaluated on the teeth, and a parental satisfaction scale will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with consenting parents,
* Patients with carious lesions on 2 or more faces of maxillary incisors or interface caries
* Those whose related teeth have not undergone pulp treatment,
* Patients without periodontal-related attachment loss, without tooth loss as a result of periodontal pathology,
* Those requiring treatment with general anaesthesia
* Score 1 and score 2 on the Frankl behaviour scale
* Those without a history of allergy (such as local anaesthesia, medication, resin-based restorative materials),
* Not requiring endocarditis prophylaxis,
* No hypoplasia and hypomineralisation of teeth,
* Patients whose permanent teeth are more than 1 year away from eruption
* Patients with vital teeth and no complaints of percussion, palpation tenderness, nocturnal waking pain and no abscess and/or fistula
* Teeth with a healthy lamina dura and periapical appearance
* Teeth without mobility and pathological gingival pockets
* Teeth with physiological root resorption not exceeding the apical 1/3 level,
* No more than 2 mm alveolar bone loss in the interproximal region on the radiograph of the tooth,
* No pathological internal or external root resorption,
* It has a permanent tooth underneath and its position is normal,
* Patients with a flush terminal closure relationship will be included in the study.

Exclusion Criteria:

* Teeth with periapical infection, abscess or mobility,
* In cases where the depth of the gingival pocket exceeds 3 mm,
* In the presence of pathological mobility,
* In the presence of congenital developmental defects (amelogenesis imperfecta, dentinogenesis imperfecta),
* In teeth in infraocclusion,
* Patients with abnormal bite due to dental or skeletal orthodontic anomalies,
* In the presence of pathological internal or external resorption,
* In cases where radiographic bone loss of more than 2 mm in the interdental region is observed
* Those with active periodontal disease,
* Traumatised teeth,
* In cases where the overjet is more than 2 mm,
* Patients with deep bite
* Cases where the opposite tooth is missing,
* Patients with systemic diseases (diseases of the cardiovascular system, endocrine system, urinary system, central nervous system, mental disorders, etc.),
* Dangerous medical conditions or harmful oral habits,
* Children with bruxism or unilateral chewing habits will not be included in the study.

Those who wish to withdraw from the study at any stage will be excluded from the study.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinical performance. | 1 week, 3 months, 6 months, 12 months
  Modified United States Public Health Service (USPHS) criteria will be used to evaluate retention, marginal integrity, secondary caries, color match, and crown fracture.
  Restorations are evaluated using an alphabetical grading scale. When assessing based on specific criteria:
  Alpha (A), represents ideal restorations, Bravo (B), denotes restorations that are not ideal but remain within acceptable limits, Charlie (C), refers to restorations that fall outside clinically acceptable boundaries and require replacement, Delta (D) is assigned to restorations that are either currently mobile or causing damage to surrounding tissues.
Change in periodontal health (Plaque) | 1 week, 3 months, 6 months, 12 months
  Periodontal health will be assessed using the Plaque index (PI).
  Each of the four surfaces of a tooth will be assigned an index score from 0 to 3 based on the amount of plaque observed:
  0: No plaque is present.
  1. A thin layer of plaque is observed along the gingival margin; this thin layer can be detected with a probe.
  2. A moderate layer of plaque is observed along the gingival margin, visible to the eye.
  3. A substantial amount of plaque is observed at the gingival margin, with interdental areas visibly filled with plaque.
Wear of opposing natural teeth | 1 week, 3 months, 6 months, 12 months
  The Smith and Knight Tooth Wear Index classification, which is used to grade tooth wear, will be applied.
  The incisal surfaces of all teeth will be examined.
  Score 0:
  (Buccal/Lingual/Occlusal/Incisal): No loss of enamel surface characteristics. (Cervical): No loss of contour.
  Score 1:
  (B/L/O/I): Loss of enamel surface characteristics. (C): Minimal loss of contour.
  Score 2:
  (B/L/O): Loss of enamel exposing dentine for less than one third of surface. (I): Loss of enamel just exposing dentine. (C): Defect less than 1 mm deep.
  Score 3:
  (B/L/O): Loss of enamel exposing dentine for more than one third of surface. (I): Loss of enamel and substantial loss of dentine (C): Defect less than 1-2 mm deep.
  Score 4:
  (B/L/O): Complete enamel loss-pulp exposure- secondary dentin exposure. (I): Pulp exposure or exposure of secondary dentine. (C): Defect more than 2 mm deep-pulp exposure- secondary dentine exposure.
Measuring of parental satisfaction | 1 week, 3 months, 6 months, 12 months
  Parental satisfaction will be evaluated on a five-point Likert scale, which responders specify their level of satisfaction.
  1. Very dissatisfied
  2. Dissatisfied
  3. Undecided
  4. Satisfied
  5. Very satisfied
Change in periodontal health (Gingiva) | 1 week, 3 months, 6 months, 12 months
  Periodontal health will be assessed using the Gingival index (GI).
  The degree of inflammation and bleeding at each of the four surfaces of a tooth will be assessed using the following index system:
  0: No visible signs of inflammation.
  1. Mild inflammation with slight color change and edema; no bleeding.
  2. Visible, moderate inflammation with a tendency to bleed when a periodontal probe is gently passed along the soft tissue wall of the gingival sulcus.
  3. Severe inflammation with marked redness, edema, and spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Görkem Ulu Güzel, Assoc. Prof., Study Director — gorkemulu@yahoo.com
Locations (1):
- Aydin Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data (IPD) will not be shared with other researchers

REFERENCES:
- [Background] Ryge G. Clinical criteria. Int Dent J. 1980 Dec;30(4):347-58. PMID 6935165
- [Background] Smith BG, Knight JK. An index for measuring the wear of teeth. Br Dent J. 1984 Jun 23;156(12):435-8. doi: 10.1038/sj.bdj.4805394. No abstract available. PMID 6590081
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Cohn C. Zirconia-Prefabricated Crowns for Pediatric Patients With Primary Dentition: Technique and Cementation for Esthetic Outcomes. Compend Contin Educ Dent. 2016 Sep;37(8):554-8. PMID 27608199
- [Background] Srinivasan SR, Mathew MG, Jayaraman J. Comparison of Three Luting Cements for Prefabricated Zirconia Crowns in Primary Molar Teeth: a 36-month Randomized Clinical Trial. Pediatr Dent. 2023 Mar 15;45(2):117-124. PMID 37106541
- [Background] Alrashdi M, Ardoin J, Liu JA. Zirconia crowns for children: A systematic review. Int J Paediatr Dent. 2022 Jan;32(1):66-81. doi: 10.1111/ipd.12793. Epub 2021 Apr 25. PMID 33772904
- [Background] Alzanbaqi SD, Alogaiel RM, Alasmari MA, Al Essa AM, Khogeer LN, Alanazi BS, Hawsah ES, Shaikh AM, Ibrahim MS. Zirconia Crowns for Primary Teeth: A Systematic Review and Meta-Analyses. Int J Environ Res Public Health. 2022 Feb 28;19(5):2838. doi: 10.3390/ijerph19052838. PMID 35270531